CLINICAL TRIAL: NCT03147053
Title: The Efficacy and Safety of Jiedu Tongluo Granules on Patients With Post-stroke Depression: a Double-blind, Randomized and Placebo-controlled Trial
Brief Title: Efficacy and Safety of Jiedu Tongluo Granules for Post-stroke Depression
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XiyuanH
Record Dates: First submitted 2017-05-01; First posted 2017-05-10 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2017-04

CONDITIONS: Post-stroke Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jiedu Tongluo granules (Experimental): Patients in this group were administered the Jiedu Tongluo granules .
  Interventions: Drug: Jiedu Tongluo granules
- Placebo (Placebo Comparator): Patients in this group were administered the placebo .
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Jiedu Tongluo granules — Patients in this group were administered the Jiedu Tongluo granules, 3.9mg/bag, 2 times/day for 8 weeks.
  Other Names: The treatment group
  Arms: Jiedu Tongluo granules
Drug: Placebo — Patients in this group were administered the placebo, 3.9mg/bag, 2 times/day for 8 weeks.
  Other Names: The control group
  Arms: Placebo

SUMMARY:
To explore the efficacy and safety of Jiedu Tongluo granules for post stroke depression. A randomized, double-blind, placebo-controlled clinical trial was designed. The treatment group was administered the Jiedu Tongluo granules, while the control group was administered the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke, with neurological deficits symptoms;
* Clinical diagnosis of depression, according to the Diagnostic and Statistical Manual of Mental Disorders-IV （DSM-IV）or Chinese Classification and Diagnostic Criteria of Mental Disorders-3(CCMD-3), the score is between 7 to 24 by 17-item Hamilton Depression;
* Age of 45 to 80 years old;
* The patient is conscious, cooperation, without aphasia and severe cognitive impairment after acute phase of stroke;
* Without psychiatric disease history or family history of psychosis before stroke;
* No hormones and psychotropic drugs were used within 1 month before enrollment;
* capacity to provide written consent.

Exclusion Criteria:

* With brain organic disease such as brain tumors;
* Had a history of psychiatric illness or depression before stroke;
* Combined with severe liver, kidney, hematopoietic system disorder;
* Poor glycemic control and insulin-dependent diabetes;
* Participate in any clinical trial or taking antidepressant treatment 1 month prior to baseline;
* Pregnant or breast feeding;
* History of sensitivity to Chinese medicine ingredients.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
Change of 17-item Hamilton Depression Scale( HAMD-17) From Baseline | 4weeks,8weeks
  Depression symptoms are mainly measured by the 17-item Hamilton Depression Scale (HAMD-17)
Change of Barthel Index (BI) From Baseline | 4weeks,8weeks
  The daily activities will be measured using Barthel Index(BI)

SECONDARY OUTCOMES:
Change of National Institute of Health stroke scale（NIHSS）From Baseline | 4weeks,8weeks
  Neurological function mainly measured by NIHSS
The stroke diagnosis and evaluation criteria of Traditional Chinese Medicine（TCM）from baseline | 4weeks,8weeks
  To evaluate patients' syndrome by TCM scale

OTHER OUTCOMES:
The change of cytokines IL-6、 IL-8 in serum from baseline | 4weeks,8weeks
  To find the inflammation factors related with post-stroke depression

CONTACTS AND LOCATIONS:
Overall Officials: Jianxun Liu, Study Director — xiyuan hospital
Locations (1):
- Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao AM, Qiu WR, Mao LJ, Ren JG, Xu L, Yao MJ, Bilinksi K, Chang D, Liu JX. The efficacy and safety of Jiedu Tongluo granules for treating post-stroke depression with qi deficiency and blood stasis syndrome: study protocol for a randomized controlled trial. Trials. 2018 May 10;19(1):275. doi: 10.1186/s13063-018-2633-4. PMID 29747670